CLINICAL TRIAL: NCT03764436
Title: Youth Leaders for Early Childhood Assuring Children Are Prepared for School - National Commission for Human Development (LEAPS-NCHD) Program Evaluation
Brief Title: LEAPS-NCHD Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Aga Khan University (Other); Yale University (Other); Swiss Tropical & Public Health Institute (Other); Dubai Cares (Other); Grand Challenges Canada (Other)
Responsible Party: Principal Investigator, Aisha K Yousafzai, Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IRB18-1149
Record Dates: First submitted 2018-11-21; First posted 2018-12-05 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Child Development
Keywords: Early Child Development; School Readiness; Early Childhood Education; Youth Development

STUDY DESIGN:
Intervention Model Description: This study uses a cluster-randomized stepped-wedge design with three steps to evaluate the impact of LEAPS-NCHD program. Ninety-nine clusters (villages) are enrolled. Thirty-three clusters per step are randomly selected to cross-over from receipt of standard services (comparison) to receipt of the LEAPS-NCHD program (intervention). Unit of randomization is at the village (cluster) level. A process evaluation will assess program rollout for fidelity, adherence, quality, and cost.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LEAPS-NCHD Program - Group 1 (Experimental): Participants will receive the LEAPS-NCHD Program, a youth-led community-based preschool program for children aged 3.5 - 5 years.
  Interventions: Behavioral: LEAPS-NCHD Program
- LEAPS-NCHD Program - Group 2 (Experimental): Participants will receive the LEAPS-NCHD Program, a youth-led community-based preschool program for children aged 3.5 - 5 years.
  Interventions: Behavioral: LEAPS-NCHD Program
- LEAPS-NCHD Program - Group 3 (Experimental): Participants will receive the LEAPS-NCHD Program, a youth-led community-based preschool program for children aged 3.5 - 5 years.
  Interventions: Behavioral: LEAPS-NCHD Program

INTERVENTIONS:
Behavioral: LEAPS-NCHD Program — The LEAPS-NCHD program trains young women aged 18 - 24 years with a minimum of 10 years of basic education to be preschool teachers, or Community Youth Leaders (CYLs) in community-based preschools in rural Sindh. CYLs will receive two weeks of classroom-based basic-training and 6 months of on-the-job coaching and support. A maximum of 20 children aged 3.5 -5 years old will be enrolled in each preschool. One preschool will be opened per cluster (village). Children will receive a minimum of 6 months of program exposure between assessment rounds.

SUMMARY:
An estimated 88 million children drop out of primary school each year worldwide, and the highest number of dropouts are in the first and second grade. A proven strategy to reduce dropout from primary school is participation in early childhood care and education (ECCE) services that bolster young children's health, development and readiness for school. Access to quality ECCE services remains highly limited in Pakistan: less than 50% of four-year-olds are estimated to attend ECCE services, and skilled ECCE workers remain scarce.

To address these challenges, LEAPS (Youth Leaders for Early Childhood Assuring Children are Prepared for School) was developed as a cross-generational strategy to support the learning and development of young children (3.5- to 5.5-year-olds) and female youth (18- to 24-year-olds). The program provides vocational training to female youth, referred to as Community Youth Leaders (CYLs), to deliver a community-based preschool program in rural Sindh, Pakistan. The LEAPS program was previously developed in partnership with Pakistan's National Commission for Human Development (NCHD), a government entity charged with supporting community health, education, and vocational training programs. Efficacy and feasibility of the LEAPS strategy were demonstrated through a prior pilot evaluated in a cluster-randomized controlled trial in 2015 (NCT02645162).

The NCHD is now seeking to integrate the LEAPS program within their full suite of services and to scale the program across 99 villages in rural Sindh under the technical guidance and support of a local implementation support team led by the Aga Khan University. This intervention utilizes two strategies: i) the first is the implementation of the LEAPS program, led by NCHD; and ii) the second is the technical support of the NCHD, to ensure the system is able to support program expansion and sustainability.

This study uses a cluster-randomized stepped-wedge design with three steps to assess program impact on school readiness and child and youth development outcomes across the 99 villages ("clusters"). All clusters will begin in the control state (i.e. access to standard community services). Prior to the start of the trial, clusters will be randomized to 'cross-over' to the intervention state (i.e. introduction of the LEAPS-NCHD program) during one of three sequential steps. Each step will be approximately 9-11 months. By the end of the trial, all clusters will have been exposed to the intervention. Measurement is assessed across all clusters at each step. The total duration of the trial will be 31 months. A process evaluation will also be conducted to examine the large-scale implementation of the LEAPS-NCHD Program.

ELIGIBILITY:
Inclusion Criteria:

* Resides in the targeted villages
* Aged 54 - 66 months
* Child's primary caregiver must provide both i) informed consent for the caregiver's own participation in the study and ii) permission for the child's participation in the study.
* Child must provide assent for participation in the study.

Exclusion Criteria:

* Child shows signs of severe clinical health condition or disability.

Ages: 54 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3858 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
School readiness | Up to 31 months
  School readiness of children aged 54 - 66 months assessed using the International Development & Early Learning Assessment (IDELA). IDELA includes domains for emergent math (7 items), socio-emotional development (5 items), self-regulation (1 item), emergent literacy (6 items), fine motor skills (3 items), and gross motor skills (1 item). Total scores are calculated for each domain, and a total IDELA score for school readiness is generated from the domain scores. Higher scores reflect better outcomes.

SECONDARY OUTCOMES:
Child executive functioning skills: working memory | Up to 31 months
  Direct assessment examining working memory capacity among children aged 54 - 66 months using the Corsi Block-tapping Test (Noel, 2009). The child's score reflects the longest sequence for which two block series were repeated correctly, plus 0.5 if one longer series was also correctly processed (range: 0 - 4 points). Higher scores indicate better outcomes.
Child general executive functioning skills | Up to 31 months
  The Head Toes Knees Shoulders task (Ponitz et al., 2008) will be used to assess general executive functioning skills among children aged 54 - 66 months. The assessment contains two sections, part one being easier and part two more challenging. Child participants may receive 0 to 20 points for each section. Scores will be presented separately for each section. Higher scores reflect better outcomes.
Child executive functioning skills: inhibitory control | Up to 31 months
  Direct assessment examining inhibitory control skills among children aged 54 - 66 months using the Knock and Tap assessment (Molfese et al., 2010). Total score is the sum across 16 items (range: 0-16 points). Higher scores reflect better outcomes.
Child executive functioning skills: inhibitory control | Up to 31 months
  Direct assessment examining inhibitory control skills among children aged 54 - 66 months using the Peg Tap assessment (range: 0-16 points) (Molfese et al., 2010). Total score is the sum across 16 items. Higher scores reflect better outcomes.
Child executive functioning skills: cognitive flexibility | Up to 31 months
  Direct assessment of cognitive flexibility skills among children aged 54 - 66 months, using the Dimensional Change Card Sort (DCCS) (Carlson, 2005). Participants are requested to sort cards at 3 levels. In the "separated" level, the cards depict a black silhouette shape (e.g., rabbit or boat) on a colored card. Thus, the shape and color dimensions are separated. In the "integrated" level, the shape and color are integrated on the card (i.e., red rabbit and blue boat). During "switch trials," participants must change the dimension being matched. In the "border" level, the integrated pictures from the previous level are used, but half of the cards have borders. Five subscores will be examined: Total number correct trials on the separated level, pre- and post-switch (0-6 points each); total number correct trials on the integrated level, pre- and post-switch (0-6 points each); and total correct on the border version (0-12 points). Higher scores reflect better outcomes.
Youth executive functioning skills: working memory | Up to 31 months
  Direct assessment to examine working memory skills of youth using the Backward Word Span task (Davis et al., 1995). The participant's score reflects the longest sequence for which two series were repeated correctly, plus 0.5 if one longer series was also correctly processed (range: 0 - 6 points). Higher scores reflect better outcomes.
Youth executive functioning skills: working memory | Up to 31 months
  Direct assessment to examine working memory capacity of youth using the Corsi Block-tapping Test (Kessels et al., 2000). Participants will be administered two tests: a forward and a backward test. A score will be awarded for each test, reflecting the longest sequence for which two series were repeated correctly, plus 0.5 if one longer series was also correctly processed (range for each: 0 - 7 points). Higher scores reflect better outcomes
Youth executive functioning skills: inhibitory control | Up to 31 months
  Direct assessment to examine inhibitory control skills of youth using the Number Stroop Effect (Stroop, 1935). Points are summed across 20 items to calculate the overall sum score (range: 0-20 points). Higher scores reflect better outcomes.
Youth executive functioning skills: cognitive flexibility | Up to 31 months
  Direct assessment to examine cognitive flexibility skills of youth using the Trail Making Task (TMT) (Lezak, 1995; Reitan & Wolfson, 1993). Scores reflect the time for completion in seconds, with the maximum time limit being 300 seconds (range: 0-300). Lower scores indicate a better outcome.
Youth personal and professional development | Up to 31 months
  Self-reported questionnaire developed for study context which includes items examining aspects of professional and personal development pertaining to autonomy, self-efficacy, self-esteem, professional growth and aspirations. This does not include a standardized scale.
Youth self-reported depressive symptoms | Up to 31 months
  Youth self-reported depressive symptoms using the Self Reporting Questionnaire 20-item (SRQ-20). Items are summed for a total score of depressive symptoms over the last 30 days (range: 0 - 20 points). Higher scores reflect poor outcomes.
Classroom structural and process quality | Assessed after program has been running for a minimum of 2 months
  Classroom quality assessed using the Measure of Early Learning Environments (MELE) module of the Measuring Early Learning Quality and Outcomes (MELQO) tool.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha K Yousafzai, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Shelina Bhamani, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Naushahro Feroze Office, Naushahro Fīroz, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on Harvard Dataverse.
Time Frame: Shared within 1 year of the end of the project; stored indefinitely on Harvard Dataverse.

REFERENCES:
- [Background] Arnold C, Bartlett K, Gowani S, Merali R. Is everybody ready? Readiness, transitions and continuity- reflections and moving forward. Working Papers in Early Childhood Development No. 41. The Netherlands: Bernard van Leer Foundation, 2007.
- [Background] UNICEF Pakistan. Out of school children in the Baluchistan, Khyber Pakhtunkhwa, Punjab and Sindh provinces of Pakistan. Islamabad: UNICEF, 2013.
- [Background] Aga Khan Foundation. Learning about Learning: Reflections on Studies from 10 Countries. Aga Khan Foundation, Geneva, Switzerland, 2013.
- [Derived] Alsager A, Franchett E, Siyal S, Bhamani S, Yousafzai AK, Sudfeld CR. Household Food Insecurity, Growth and Development of Preschool Children: Evidence From Rural Pakistan. Matern Child Nutr. 2025 Oct;21(4):e70062. doi: 10.1111/mcn.70062. Epub 2025 Jul 7. PMID 40621881
- [Derived] Yousafzai AK, Siyal S, Franchett EE, Dai Q, Rehmani K, Sudfeld CR, Bhamani S, Hakro S, Reyes CR, Fink G, Ponguta LA. Effect of a youth-led early childhood care and education programme on children's development and learning in rural Sindh, Pakistan (LEAPS): a stepped-wedge cluster-randomised implementation trial. Lancet Child Adolesc Health. 2025 Jan;9(1):25-36. doi: 10.1016/S2352-4642(24)00304-3. Epub 2024 Dec 2. PMID 39637878
- [Derived] Ali NB, Yousafzai AK, Siyal S, Bhamani S, Sudfeld CR. Effect of a Center-Based Early Childhood Care and Education Program on Child Nutritional Status: A Secondary Analysis of a Stepped-Wedge Cluster Randomized Controlled Trial in Rural Sindh, Pakistan. J Nutr. 2024 Feb;154(2):755-764. doi: 10.1016/j.tjnut.2023.12.008. Epub 2023 Dec 9. PMID 38072156
- [Derived] Yousafzai AK, Sudfeld CR, Franchett EE, Siyal S, Rehmani K, Bhamani S, Dai Q, Reyes CR, Fink G, Ponguta LA. Evaluating implementation of LEAPS, a youth-led early childhood care and education intervention in rural Pakistan: protocol for a stepped wedge cluster-randomized trial. Trials. 2021 Aug 17;22(1):542. doi: 10.1186/s13063-021-05518-9. PMID 34404454